CLINICAL TRIAL: NCT05046652
Title: Effectiveness of Convalescent Plasma Therapy in 8 Non-Intubated COVID-19 Patients in Indonesia: A Case Series
Status: Completed | Type: Observational
Sponsor: Maranatha Christian University (Other)
Collaborators: Primaya Hospital Tangerang Indonesia (Unknown)
Responsible Party: Principal Investigator, Theresia Monica Rahardjo, Director of Unggul Karsa Medika Hospital, Maranatha Christian University
Other Study IDs: 0408087106
Record Dates: First submitted 2021-04-12; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Infectious Disease
Keywords: convalescent plasma therapy; non-intubated; case studies; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Communicable Diseases; COVID-19 | interventions — Immunization, Passive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- One bag of convalescent plasma therapy: Four patients had been administered one dose of 200 mL CP with an antibody titer of 1:320.
  Interventions: Biological: Convalescent Plasma Therapy
- Two bags of convalescent plasma therapy: Four patients had been administered two doses of 200 mL CP with an antibody titer of 1:320.
  Interventions: Biological: Convalescent Plasma Therapy

INTERVENTIONS:
Biological: Convalescent Plasma Therapy — In this study, eight non-intubated Covid-19 patients confirmed by real-time viral RNA PCR tests were included. Four patients had been administered two doses of 200 mL convalescent plasma (CP) and another four patients had been administered one dose of CP with an antibody titer of 1:320.

SUMMARY:
This is the first Case Studies article highlight factors determine the effectiveness of Convalescent Plasma Therapy (CPT) in Indonesia, accompanied by supporting data and images before and after the patients received the therapy. This Case Studies gives a huge contribution as CPT still on going as multicentre study and apply massively as emergency approved treatment in Indonesia.

DETAILED DESCRIPTION:
Eight non-intubated Covid-19 patients confirmed by real-time viral RNA PCR tests were included. Four patients had been administered two doses of 200 mL convalescent plasma (CP) and another four patients had been administered one dose of CP with an antibody titer of 1:320. This study has three goals included to detect the improvement of patient clinical and laboratory conditions, safety of CPT, and conversion from positive to negative results after CPT administration. Convalescent plasma applied within two weeks (13 days) from onset of illness and within a week (6.5 days) from the first day of hospital admission for all patients. Improvements in clinical symptoms, laboratory parameters, thorax photo, negative conversion of PCR, and decreased oxygen supplementation occurred within a week after CPT. Patients with two doses of CP tended to have faster recovery than those with one dose of CP. No severe adverse effects were observed in any patient. This is the first case series in Indonesia showing CPT is safe and well tolerated, and early CPT before the patient is intubated could potentially prevent disease progression, increase the recovery rate, and shorten the inpatient days.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients
* Severe stage
* Positive PCR swab

Exclusion Criteria:

* Non-COVID-19 patients
* No Symptoms COVID-19 patients
* Mild COVID-19 patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eight patients originated from one region of Tangerang with positive PCR swab
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Patients with two doses of CP tended to have faster recovery than those with one dose of CP. | 1 April 2020 - 31 December 2020
  The median time from onset of illness to CPT was 13 days (within two weeks), and from the first day of hospital admission to CPT was 6.5 days (within a week). There were improvements in clinical symptoms, laboratory parameters, thorax photo, negative conversion of PCR, and decreased oxygen supplementation within a week after CPT. No severe adverse effects were observed in any patient.

SECONDARY OUTCOMES:
Patients with two doses of CP tended to have faster PCR negative conversion time than those with one dose of CP | 1 April 2020 - 31 December 2020
  All four patients given two doses of CP became negative in PCR swab but only two of four patients given one dose of CPT showed negative PCR swab result

CONTACTS AND LOCATIONS:
Overall Officials: Theresia M Rahardjo, Dr, Principal Investigator — Maranatha Christian University
Locations (1):
- Theresia Monica Monica, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Indonesia: WHO Coronavirus Disease (COVID-19) Dashboard | WHO Coronavirus Disease (COVID-19) Dashboard
- [Background] Ozdemir OHE. Convalescent (Immune) Plasma Therapy with all Aspects: Yesterday, Today and COVID-19. Erciyes Med J. 2020;1-8.
- [Background] Rahardjo TM, Triyono T, Harly PR. Buku Penatalaksanaan Terapi Plasma Konvalesen Bagi Pasien COVID-19 Di Indonesia. Revised Edition. September 2020.
- [Result] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Result] Focosi D, Anderson AO, Tang JW, Tuccori M. Convalescent Plasma Therapy for COVID-19: State of the Art. Clin Microbiol Rev. 2020 Aug 12;33(4):e00072-20. doi: 10.1128/CMR.00072-20. Print 2020 Sep 16. PMID 32792417
- [Result] Bloch EM, Shoham S, Casadevall A, Sachais BS, Shaz B, Winters JL, van Buskirk C, Grossman BJ, Joyner M, Henderson JP, Pekosz A, Lau B, Wesolowski A, Katz L, Shan H, Auwaerter PG, Thomas D, Sullivan DJ, Paneth N, Gehrie E, Spitalnik S, Hod EA, Pollack L, Nicholson WT, Pirofski LA, Bailey JA, Tobian AA. Deployment of convalescent plasma for the prevention and treatment of COVID-19. J Clin Invest. 2020 Jun 1;130(6):2757-2765. doi: 10.1172/JCI138745. PMID 32254064
- [Result] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Result] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Result] Abolghasemi H, Eshghi P, Cheraghali AM, Imani Fooladi AA, Bolouki Moghaddam F, Imanizadeh S, Moeini Maleki M, Ranjkesh M, Rezapour M, Bahramifar A, Einollahi B, Hosseini MJ, Jafari NJ, Nikpouraghdam M, Sadri N, Tazik M, Sali S, Okati S, Askari E, Tabarsi P, Aslani J, Sharifipour E, Jarahzadeh MH, Khodakarim N, Salesi M, Jafari R, Shahverdi S. Clinical efficacy of convalescent plasma for treatment of COVID-19 infections: Results of a multicenter clinical study. Transfus Apher Sci. 2020 Oct;59(5):102875. doi: 10.1016/j.transci.2020.102875. Epub 2020 Jul 15. PMID 32694043
- [Result] Liu STH, Lin HM, Baine I, Wajnberg A, Gumprecht JP, Rahman F, Rodriguez D, Tandon P, Bassily-Marcus A, Bander J, Sanky C, Dupper A, Zheng A, Nguyen FT, Amanat F, Stadlbauer D, Altman DR, Chen BK, Krammer F, Mendu DR, Firpo-Betancourt A, Levin MA, Bagiella E, Casadevall A, Cordon-Cardo C, Jhang JS, Arinsburg SA, Reich DL, Aberg JA, Bouvier NM. Convalescent plasma treatment of severe COVID-19: a propensity score-matched control study. Nat Med. 2020 Nov;26(11):1708-1713. doi: 10.1038/s41591-020-1088-9. Epub 2020 Sep 15. PMID 32934372
- [Result] Libster R, Perez Marc G, Wappner D, Coviello S, Bianchi A, Braem V, Esteban I, Caballero MT, Wood C, Berrueta M, Rondan A, Lescano G, Cruz P, Ritou Y, Fernandez Vina V, Alvarez Paggi D, Esperante S, Ferreti A, Ofman G, Ciganda A, Rodriguez R, Lantos J, Valentini R, Itcovici N, Hintze A, Oyarvide ML, Etchegaray C, Neira A, Name I, Alfonso J, Lopez Castelo R, Caruso G, Rapelius S, Alvez F, Etchenique F, Dimase F, Alvarez D, Aranda SS, Sanchez Yanotti C, De Luca J, Jares Baglivo S, Laudanno S, Nowogrodzki F, Larrea R, Silveyra M, Leberzstein G, Debonis A, Molinos J, Gonzalez M, Perez E, Kreplak N, Pastor Arguello S, Gibbons L, Althabe F, Bergel E, Polack FP; Fundacion INFANT-COVID-19 Group. Early High-Titer Plasma Therapy to Prevent Severe Covid-19 in Older Adults. N Engl J Med. 2021 Feb 18;384(7):610-618. doi: 10.1056/NEJMoa2033700. Epub 2021 Jan 6. PMID 33406353
- [Result] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Result] Sun M, Xu Y, He H, Zhang L, Wang X, Qiu Q, Sun C, Guo Y, Qiu S, Ma K. A potentially effective treatment for COVID-19: A systematic review and meta-analysis of convalescent plasma therapy in treating severe infectious disease. Int J Infect Dis. 2020 Sep;98:334-346. doi: 10.1016/j.ijid.2020.06.107. Epub 2020 Jul 4. PMID 32634589
- [Result] Cao WC, Liu W, Zhang PH, Zhang F, Richardus JH. Disappearance of antibodies to SARS-associated coronavirus after recovery. N Engl J Med. 2007 Sep 13;357(11):1162-3. doi: 10.1056/NEJMc070348. No abstract available. PMID 17855683
- [Result] Aviani JK, Halim D, Soeroto AY, Achmad TH, Djuwantono T. Current views on the potentials of convalescent plasma therapy (CPT) as Coronavirus disease 2019 (COVID-19) treatment: A systematic review and meta-analysis based on recent studies and previous respiratory pandemics. Rev Med Virol. 2021 Nov;31(6):e2225. doi: 10.1002/rmv.2225. Epub 2021 Feb 23. PMID 33621405